CLINICAL TRIAL: NCT02842775
Title: Clinical Evaluation and Rehabilitation System for Dynamic Balance Control in Cervical Myelopathy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201512167RINB
Record Dates: First submitted 2016-07-11; First posted 2016-07-25 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2019-04

CONDITIONS: Cervical Myelopathy
Keywords: rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dynamic balance exercise group (Experimental): balance perturbation training
  Interventions: Other: balance perturbation training
- Control group (No Intervention): No intervention

INTERVENTIONS:
Other: balance perturbation training — perturbation training on the split-belt balance perturbance treadmill,
  Arms: Dynamic balance exercise group

SUMMARY:
Cervical myelopathy is common among the aging population.One of the complications of cervical myelopathy is balance impairment.In this study, the patients with cervical myelopathy undergo biomechanical, imaging, neurophysiological and functional assessment. Besides, the dynamic balance training is introduced to the patients with cervical decompression surgery.This study is expected to provide important empirical evidence to evaluate the prognosis of the surgery, to further guide the postoperative rehabilitation of myelopathy patients and to improve patients' long-term quality of life.

DETAILED DESCRIPTION:
Taiwan is quickly becoming a nation of the aging population with myelopathy reporting to be one of the most common spinal cord disorders associated with spinal degeneration. Given the high prevalence rate of the condition, current project aims to investigate the impact of myelopathy on motor control from a biomechanical perspective with the overall aim to develop an interactive balance perturbation rehabilitation program targeting individual patients and identified the deficiency. The efficacy of the individual rehabilitation program will be assessed and determined to utilize a prospective longitudinal study design. A break down of the proposed three-year project are as follows:

Year 1: Myelopathy patients prepared to receive cervical decompression surgery as well as age-matched asymptomatic controls will be recruited and subjected to the following clinical evaluations: 3-dimensional biomechanical motion analysis, diagnostic Magnetic Resonance Imaging, pain and disability questionnaires, motor performance assessment, spinal curvature, muscle strength assessment as well as transcranial magnetic stimulation examination. Motor control and coordination of functional movements will also be evaluated.

Year 2: Continue to recruit potential participants and further develop the use of the interactive split-belt balance perturbation treadmill as modalities for gait and balance therapy.

Year 3: Physical Therapy rehabilitation programs at 3-month post surgery, one group will participate in a specific and personalized interactive balance perturbation training program targeting balance and gait retraining, while the other group receives the routine Physical Therapy program. Both treatment groups will be assessed pre-operatively, at 3, 6 and 12 months postoperatively. Patients will be classified based on their severity and grade of the spinal cord compression before being compared for any difference in treatment responses.

Year 4: Follow-up monitoring and documenting the number of falls experienced by patients at one year postoperatively as an outcome of effectiveness.

Expected outcome and significance The findings from the current project will provide important empirical evidence to guide the postoperative rehabilitation of myelopathy patients. Through detailed biomechanical motion analysis, it is anticipated that this project will provide an in-depth understanding of the influence of decompression surgery on motor control and spinal stability. The tailored and innovative rehabilitation program will also improve patients' long-term quality of life.

ELIGIBILITY:
Inclusion criteria:

* Aged 40-80 years old
* Diagnosed cervical myelopathy according MRI imaging
* Able to stand more than 30 seconds

Exclusion criteria:

* With rheumatoid arthritis, ankylosing spondylitis,multiple sclerosis and other systemic disorders
* With musculoskeletal or neurological disorders,which can impair balance
* With previous spinal surgery
* Unable to communicate or follow instruction
* Not suit to cervical decompressive surgery or physical therapy due to other medical condition

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-01; Primary Completion 2018-01-22 (Actual); Study Completion 2018-01-22 (Actual)

PRIMARY OUTCOMES:
Kinematics (joint range of motion) | 1 year
  joint range of motion
Electromyography(EMG) | 1 years
  EMG of lower extremity
Muscle Strength Assessment by Dynamometer | 1 years
  Muscle strength of upper and lower extremity
Kinetic(Ground reaction force) | 1 years
  Ground reaction force
Transcranial magnetic stimulation (TMS) | 1 years

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | 3 years
Neck Disability Index (NDI) | 3 years
Japanese Orthopaedic Association Myelopathy Evaluation Questionnaire(JOACMEQ) | 3 years
Nurick Classification | 3 years
Five Times Sit to Stand Test | 3 years
Timed Up & Go test (TUG) | 3 years
Dynamic Gait Index (DGI) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Li Hsu, Principal Investigator — School and Graduate Institute of Physical Therapy, College of Medicine,National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan